CLINICAL TRIAL: NCT05488249
Title: CCTA Study of Atheromatous Lesions, Coronary Hemodynamics and Systemic Inflammation in Patients With Vulnerable Plaques (COHESIVE STUDY)
Brief Title: CCTA Coronary Hemodynamics, Systemic Inflammation and Vulnerable Plaques (COHESIVE)
Acronym: COHESIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM-75/2022-COHESIVE
Record Dates: First submitted 2022-07-30; First posted 2022-08-04 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease; Systemic Inflammatory Response; Chronic Coronary Syndrome; Atherosclerosis
Keywords: coronary vulnerable plaque; CCTA; Systemic inflammation; Coronary shear stress; Plaque topography
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood sampling during CCTA image acquisition for evaluation of systemic inflammation (based on hsCRP, interleukin-6, MMP-9, V-CAM, I-CAM, e-selectin, p-selectin, periostin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac imaging tests — * 2D transthoracic echocardiography
  * 128-multislice CT coronary angiography with the evaluation of: epicardial fat volume, plaque burden, total and local calcium score, markers for lesion severity; morphological plaque characteristics; plaque components evaluated via volumetric and planimetric units; markers of plaque vulnerability (necrotic core, low attenuation plaque, spotty calcification, napkin ring sign, positive remodeling).
  * Shear stress evaluation via computational fluid dynamics.
Diagnostic Test: Venous blood sample collection — Venous blood sample collection during CCTA image acquisition for evaluation of serum levels of hsCRP, IL-6, matrix metalloproteases - MMP9, Adhesion molecules (VCAM, ICAM, e-selectin, p-selectin) periostin.

SUMMARY:
Although there are numerous studies that have demonstrated the impact of systemic inflammation on coronary plaque vulnerability, there are few literature data regarding the influence of coronary plaque localization within the coronary tree (right and left coronary artery, proximal, mid-coronary and distal), on plaque composition, morphology and degree of vulnerability, in relation with systemic inflammation and coronary hemodynamics. The aim of this study is to identify: (1) the impact of plaque topography in different sites within the coronary tree (right versus left, proximal distal) on their vulnerability degree evaluated with CCTA; (2) the relationship between degree of plaque vulnerability, systemic inflammatory biomarkers and specific hemodynamic characteristics quantified by coronary shear stress computations. The study will include 100 patients with stable coronary artery disease for which data collection will be perform on: (1) Clinical, echocardiographic and ECG data; (2) cardiovascular risk assessment; (3) 128 slice CCTA evaluation of coronary tree anatomy, plaque morphology, composition and vulnerability degree; (4) systemic inflammation based on serum levels of hsCRP, IL-6, MMP-9, periostin, adhesion molecules (5) shear stress via coronary flow computational simulations.

DETAILED DESCRIPTION:
This is a clinical, observational cross sectional, mono-centric study which will be carried out in the Center of Advanced Research in Multimodal Cardiac Imaging Cardiomed in collaboration with the University of Medicine, Pharmacy, Sciences and Technology "GE Palade".

The project will include 100 subjects with stable coronary artery disease (defined according to the ESC guidelines for management of patients with chronic coronary syndromes), presenting in out-patient conditions, who will undergo 128 slice CCTA evaluation of coronary artery tree anatomy, coronary plaque morphology, composition and degree of vulnerability.

Samples for systemic serum biomarkers for systemic inflammation will be collected at the moment of CCTA image acquisition for all patients. The endothelial coronary shear stress will be calculated with imaging post-processing techniques on the CT data acquired at baseline, by using computational fluid dynamics.

The study will be conducted over a period of 6 months, in which patients will be examined for clinical data, echocardiography assessment of left ventricular function, valvular disease, diastolic function, 12-lead ECG, cardiovascular risk assessment, systemic inflammation (based on serum levels of hsCRP, interleukin-6, MMP-9, periostin, adhesion molecules. Coronary plaque analysis will be conducted on an offline station by using dedicated post-processing software for detection of plaque morphology (length, volume, degree of stenosis, plaque location within the coronary tree, remodeling and eccentricity index), composition (lipid rich, fibrotic and calcified volumes), degree of vulnerability (identification of positive remodeling, low attenuation, spotty calcium, napkin ring sing). After plaque selection and analysis, computational fluid dynamics based on CCTA images will be performed on an offline dedicated station for coronary shear stress quantification.

Primary exclusion criteria include acute coronary syndromes at the moment of enrollment, with myocardial necrosis, the presence of coronary stents and extensive calcifications and suboptimal CCTA image acquisition that could interfere with plaque analysis, as well as contraindications for administration of contrast media agent (renal disease, allergies, thyroid dysfunction).

Study objectives:

Primary: to investigate the association between coronary plaque topography in different sites within the coronary tree (right versus left, proximal distal) and their vulnerability degree evaluated with CCTA.

Secondary: to assess the relationship between degree of plaque vulnerability, systemic inflammatory biomarkers and specific hemodynamic characteristics quantified by coronary shear stress computations in relation to plaque location.

Study procedures

* Clinical examination, medical history, cardiovascular risk assessment
* 12-lead ECG
* 2D transthoracic echocardiography with measurement of: cardiac diameters, volumes, valvular function and regurgitation, pressure gradients, pericardial fat thickness, pericardial effusion, left ventricular global and regional function and ejection fraction.
* 128-multislice CT coronary angiography with the evaluation of: epicardial fat volume, plaque burden, total and local calcium score, markers for lesion severity (degree of stenosis, lesion length, lumen area and diameter, minimum and maximum plaque thickness); morphological plaque characteristics (plaque related volumes, plaque burden, vascular indexes - remodeling and eccentricity index); plaque components evaluated via volumetric and planimetric units (necrotic core, fibrofatty tissue, fibrotic tissue, dense calcium); markers of plaque vulnerability (necrotic core, low attenuation plaque, spotty calcification, napkin ring sign, positive remodeling).
* Shear stress evaluation of CT acquired images and computational fluid dynamics
* Venous blood sample collection during the acute coronary event for evaluation of serum levels of hsCRP, IL-6, matrix metalloproteases - MMP9, Adhesion molecules (VCAM, ICAM, e-selectin, p-selectin), periostin.
* Data collection: In a dedicated database that includes all patient information, demographics, medical history, medication, therapeutic procedures, information derived from imaging techniques (echocardiography, CT angiography, CT imaging post-processing and shear stress evaluation).

ELIGIBILITY:
Inclusion Criteria:

* chronic coronary syndromes (defined according to current ESC guidelines) presenting in out-patient conditions for CCTA evaluation of stable chest pain
* age over 30 years

Exclusion Criteria:

* the presence of acute coronary syndromes at the moment of enrollment
* the presence of coronary stents and severe calcifications or other conditions that could interfere with image postprocessing and coronary plaque analysis
* acute renal failure of end-stage chronic kidney disease
* contraindication for iodine contrast agent administration (allergies, thyroid dysfunction, etc)
* active malignancy or history of cancer within the last 12 months prior to enrollment.
* systemic inflammatory disease, acute infections, positive SARS-CoV2 test, or other conditions that could interfere with the systemic inflammatory response.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable chest pain who present in out-patient conditions for complete clinical assessment and CCTA evaluation of coronary artery tree, without any history of coronary revascularization, with a low to intermediate pre-test probability for coronary artery disease, who do not present acute or chronic inflammatory/infections disease or malignancy that could interfere with the systemic inflammatory response.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Relationship between coronary plaque localization on its degree of vulnerability | through study completion, an average of 1 year
  Calculating correlations between analyzed lesion topography (right versus left coronary artery, proximal versus distal vascular localization) and indicators of plaque morphology *(volume, length, degree of stenosis), plaque composition (calcified, fibrotic, lipid rich volumes), and degree of vulnerability (quantified by the presence of low attenuation plaque, spotty calcium, napkin ring sign, positive remodeling, number of vulnerability markers)

SECONDARY OUTCOMES:
Relationship between systemic inflammation on coronary plaque vulnerability, according to plaque location and hemodynamic characteristics | through study completion, an average of 1 year
  Evaluation of association between serum levels of inflammatory biomarkers (hsCRP, IL-6, MMP-9, V-CAM, I-CAM, selectins, periostin) and markers of plaque characterization (morphology, composition degree of vulnerability) in relation to the coronary hemodynamic characteristics (by quantification of coronary shear stress based on CCTA images).

CONTACTS AND LOCATIONS:
Overall Officials: Diana Opincariu, MD, PhD, Study Director — CardioMed Medical Center
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Romania

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available for interested parties.
Supporting Information: Study Protocol
Time Frame: The IPD sharing frame is starting 6 months after publication.

REFERENCES:
- [Background] Opincariu D, Benedek T, Chitu M, Rat N, Benedek I. From CT to artificial intelligence for complex assessment of plaque-associated risk. Int J Cardiovasc Imaging. 2020 Dec;36(12):2403-2427. doi: 10.1007/s10554-020-01926-1. Epub 2020 Jul 2. PMID 32617720
- [Background] Opincariu D, Rodean I, Rat N, Hodas R, Benedek I, Benedek T. Systemic Vulnerability, as Expressed by I-CAM and MMP-9 at Presentation, Predicts One Year Outcomes in Patients with Acute Myocardial Infarction-Insights from the VIP Clinical Study. J Clin Med. 2021 Jul 31;10(15):3435. doi: 10.3390/jcm10153435. PMID 34362217
- [Background] Mester A, Rat N, Benedek T, Opincariu D, Hodas R, Chitu M, Benedek I. Acute-Phase Inflammatory Reaction Predicts CMR Myocardial Scar Pattern and 2-Year Mortality in STEMI Patients Undergoing Primary PCI. J Clin Med. 2022 Feb 24;11(5):1222. doi: 10.3390/jcm11051222. PMID 35268316
- [Background] Opincariu D, Rat N, Mester A, et al. Site-specific Phenotype of Atherosclerotic Lesions According to Their Location Within the Coronary Tree - a CCTA-based Study of Vulnerable Plaques. Journal of Cardiovascular Emergencies 2021;7(2):39-46. DOI: 10.2478/jce-2021-0010
- [Background] DISCHARGE Trial Group; Maurovich-Horvat P, Bosserdt M, Kofoed KF, Rieckmann N, Benedek T, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Cemerlic Adic N, Gutberlet M, Dodd JD, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Kubiak C, Gutierrez-Ibarluzea I, Schultz Hansen K, Muller-Nordhorn J, Merkely B, Knudsen AD, Benedek I, Orr C, Xavier Valente F, Zvaigzne L, Suchanek V, Zajanckauskiene L, Adic F, Woinke M, Hensey M, Lecumberri I, Thwaite E, Laule M, Kruk M, Neskovic AN, Mancone M, Kusmierz D, Feuchtner G, Pietila M, Gama Ribeiro V, Drosch T, Delles C, Matta G, Fisher M, Szilveszter B, Larsen L, Ratiu M, Kelly S, Garcia Del Blanco B, Rubio A, Drobni ZD, Jurlander B, Rodean I, Regan S, Cuellar Calabria H, Boussoussou M, Engstrom T, Hodas R, Napp AE, Haase R, Feger S, Serna-Higuita LM, Neumann K, Dreger H, Rief M, Wieske V, Estrella M, Martus P, Dewey M. CT or Invasive Coronary Angiography in Stable Chest Pain. N Engl J Med. 2022 Apr 28;386(17):1591-1602. doi: 10.1056/NEJMoa2200963. Epub 2022 Mar 4. PMID 35240010
- [Background] Szilveszter B, Celeng C, Maurovich-Horvat P. Plaque assessment by coronary CT. Int J Cardiovasc Imaging. 2016 Jan;32(1):161-72. doi: 10.1007/s10554-015-0741-8. Epub 2015 Aug 18. PMID 26280890